CLINICAL TRIAL: NCT04164953
Title: Tolerance and Efficacy Study of Second-line Surgery After Percutaneous Needle Aponeurotomy for Dupuytren's Disease. URAM 3
Brief Title: Tolerance and Efficacy Study of Second-line Surgery After Percutaneous Needle Aponeurotomy for Dupuytren's Disease.
Acronym: URAM3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr ROULOT (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A03363-50
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-09

CONDITIONS: Dupuytren's Disease; Surgical Incision
MeSH Terms: conditions — Dupuytren Contracture; Surgical Wound | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Surgical intervention as second-line surgery for the treatment of Dupuytren's disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dupuytren's (Experimental): Surgical intervention as second-line surgery for the treatment of Dupuytren's disease.
  Interventions: Procedure: Surgical treatment

INTERVENTIONS:
Procedure: Surgical treatment — Surgical treatment of Dupuytren's disease. Average from 2 to 4 joints per hand operated on simultaneously

SUMMARY:
As part of a graduated medical-surgical strategy, and in our practice, surgery for Dupuytren's disease appears as a second-line treatment indicated in a situation of failure after treatment with percutaneous needle aponeurotomy.The results of second-line surgery in terms of safety and efficacy have not been specifically evaluated in patients who underwent failed percutaneous needle aponeurotomy. This evaluation nevertheless appears necessary for the validation of a medical-surgical strategy during Dupuytren's disease.

DETAILED DESCRIPTION:
Dupuytren's disease is characterised by retractile fibrosis of the superficial palmar aponeurosis that can result in irreversible flexing of the fingers and long-term disability. The treatment of Dupuytren's disease, whether medical or surgical, remains symptomatic. It is based in Europe on percutaneous needle aponeurotomy and surgical aponeurectomy. Its objectives are the reduction of the deformity of the fingers in flexum, and that of the incapacity that generates the illness. Percutaneous needle aponeurotomy for Dupuytren's disease was developed by Jean-Luc Lermusiaux in 1972 in the Rheumatology Department of the Lariboisière Hospital in Paris. Its efficiency, its tolerance, its simplicity, its low cost and the possibility of repeating it make it a benchmark treatment. Percutaneous needle aponeurotomy is, for many, if the existence of this technique is known and understood, the first-line treatment of Dupuytren's disease.

As part of a graduated medical-surgical strategy, and in our practice, surgery for Dupuytren's disease appears as a second-line treatment indicated in a situation of failure after treatment with percutaneous needle aponeurotomy. The safety and efficacy of the surgery was evaluated in the context of a first-line treatment of Dupuytren's disease. The results of second-line surgery in terms of safety and efficacy have not been specifically evaluated in patients who underwent failed percutaneous needle aponeurotomy. This evaluation nevertheless appears necessary for the validation of a medical-surgical strategy during Dupuytren's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Dupuytren's disease previously treated by percutaneous needle aponeurotomy and not satisfied after a delay of at least one month in regards to at least one of the treated segments (are you satisfied? response no)
* Keeping a flexum > 20°
* At least 18 years old
* Informed about the study and having given their informed and written consent for participation
* Registered with a social security scheme or the CMU (beneficiary or entitled)
* having had a medical examination confirming the surgical indication (the results of which were communicated to them).

Exclusion Criteria:

* Cognitive disorders deemed incompatible with participation in the trial by the researcher (inability to understand the information, give informed consent or follow the required assessments)
* Pregnancy in progress confirmed by interview
* language barrier that would prevent the achievement of a reliable evaluation
* Superficial or deep palmo-digital infection or inflammation
* Ruptured tendon of the flexor digitorum
* Contraindication to surgery or anaesthesia
* Participation of the patient in another clinical study in progress.
* Protected adults under guardianship, trusteeship or other legal protection, deprived of liberty by judicial or administrative decision, Pregnant, lactating or parturient women, Hospitalised without consent.

  9- Patient who has already undergone the surgical procedure under study on one of the two hands in the last 12 months or patient requiring surgery for the second hand in the next 14 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2020-06-05 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
joint deformity | 3 months
  Primary end point: joint deformity of each treated joint at 3 months.• The development of the degree of joint extension malalignment at 3 months will be described both by the relative difference and by the absolute difference between the measurements at V0 and V3, overall and for each modality of the known prognostic factors: joint types (MCP versus PIP), age at onset of disease (<50 years versus >= 50 years), initial severity of disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic Jouvenet, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: Undecided